CLINICAL TRIAL: NCT00486694
Title: A Randomised Non-Inferiority Trial of Sulfadoxine-Pyrimethamine Plus Artesunate Compared to Chloroquine for the Treatment of Vivax Malaria in Eastern Afghanistan.
Brief Title: Artesunate Plus Sulfadoxine-Pyrimethamine Versus Chloroquine for Vivax Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T26/181/33
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2007-06-15 (Estimated); Status verified 2007-06

CONDITIONS: Malaria, Vivax
Keywords: Malaria, vivax; Afghanistan; Sulfadoxine-pyrimethamine; drug resistance
MeSH Terms: conditions — Malaria, Vivax | interventions — sulfadoxine-pyrimethamine-artesunate; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine + artesunate
Drug: Chloroquine

SUMMARY:
The purpose of this study was to determine whether the proposed first line treatment for falciparum malaria in this region (sulfadoxine-pyrimethamine + artesunate) would be no worse a treatment for vivax malaria that the standard vivax treatment of chloroquine. In areas where vivax and falciparum malaria co-exist misdiagnosis of vivax malaria as falciparum is not unlikely; it is important to know whether adequate treatment will be received in these cases.

DETAILED DESCRIPTION:
In areas co-endemic for falciparum and vivax malaria incorrect differential diagnosis is always a risk. Where the recommended treatment for the two diseases is the same this presents no problem for effective treatment or clinical cure of either species. Chloroquine remains an effective treatment of choice for vivax malaria in most settings, but with the spread of chloroquine-resistant falciparum malaria across Asia, many countries now use artemisinin-based combination therapy for this species of malaria. Differential diagnostic practices, have not improved in parallel. In Afghanistan the adoption of sulfadoxine-pyrimethamine plus artesunate (SP+AS) as first-line falciparum treatment raises the prospect of a significant proportion of vivax malaria being misdiagnosed and treated with the combination. SP is considered to have limited efficacy against vivax malaria and the efficacy of SP+AS against vivax has not been established in areas that have made the switch. A randomized, non-inferiority trial comparing SP+AS (1 day SP, 3 days AS) to chloroquine monotherapy was undertaken on 190 vivax patients in Eastern Afghanistan. A margin of equivalence of 14%, with 90% power and 95% CI (two-sided α = 0.05) was used. Standard WHO procedures for in vivo evaluation of antimalarial drugs were followed. 180 individuals completed the trial to day 42. The primary outcome was proportion of patients free from failure at day 28. Using a per protocol analysis both regimens resulted in ≥96% treatment success at 28 days, but significantly more cases failed in the CQ arm (46%) than in the SP+AS arm (24%) by day 42. Based on predetermined statistical criteria SP+AS was shown to be non-inferior to the standard chloroquine treatment. In areas where vivax infections might be misdiagnosed as falciparum infections and treated with SP+AS, patient management would be as good or better than with the standard CQ treatment.

ELIGIBILITY:
Inclusion Criteria:

* microscopy confirmed P. vivax mono-infection
* age >2 years
* weight >5kg
* >1 asexual parasite per 10 fields

Exclusion Criteria:

* pregnant
* evidence of concomitant infection or serious disease
* recent use of antimalarial drugs
* severe malaria
* known allergy to study drugs

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2004-03; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with parasitological cure up to day 28 after treatment (defined as clearance of circulating vivax parasites by day 7 and absence until end of follow-up).

SECONDARY OUTCOMES:
Parasite and fever clearance times, the proportion of patients free of parasites at 42 days, and the proportion of patients with detectable gametocytes during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Rowland, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine

REFERENCES:
- [Derived] Kolaczinski K, Durrani N, Rahim S, Rowland M. Sulfadoxine-pyrimethamine plus artesunate compared with chloroquine for the treatment of vivax malaria in areas co-endemic for Plasmodium falciparum and P. vivax: a randomised non-inferiority trial in eastern Afghanistan. Trans R Soc Trop Med Hyg. 2007 Nov;101(11):1081-7. doi: 10.1016/j.trstmh.2007.06.015. Epub 2007 Aug 17. PMID 17707447